CLINICAL TRIAL: NCT03246204
Title: Chinese Observational Prospective Study of Aging Population With Chronic Kidney Disease(C-OPTION)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Fudan University (Other); China-Japan Friendship Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); Shandong Provincial Hospital (Other Government); Beijing Friendship Hospital (Other); RenJi Hospital (Other); Hebei Medical University Third Hospital (Other); Second Hospital of Jilin University (Other); Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Chen Xiangmei, Academician of Chinese Academy of Engineering, Chinese PLA General Hospital
Other Study IDs: 2015BAI12B06
Record Dates: First submitted 2017-06-13; First posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, whole blood，urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is an observational, multicenter, prospective cohort study aimed at evaluating a 5-year screening programme for chronic kidney disease(CKD) in a population of elderly patients, aged 65 years or more, in China.To analyze the etiology and composition spectrum, the incidence of complications and co-morbidities.To assess the correlation between daily living ability, mental and physical function, quality of life, nutritional status and prognosis.To develop biomarkers of renal aging.

ELIGIBILITY:
Inclusion Criteria:

* age≥65 years
* clinical diagnosis of CKD
* signed informed consent

Exclusion Criteria:

* subjects who have a poor compliance and cannot be scheduled for follow-up
* subjects participating in other interventional clinical trials
* ESRD or dialysis
* Acute kidney injury(AKI)
* history of solid organ or bone marrow transplantation
* active malignancy within 24 months prior to screening or metastatic cancer
* life expectancy less than 6 months；
* severe cognitive impairment（NYHA III or IV）
* HIV infection or AIDS
* subjects cannot be able to complete the assessment including dementia or other mental disorders, limited physical activity, severe visual impairment
* simple hematuria

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: subjects with 65 years or older
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Death | 5 year
Incidence of End Stage Renal Disease (ESRD) | 5 year
  ESRD will be defined as estimated glomerular filtration rate(eGFR)<15 mL/min/1.73 m2 or dialysis
eGFR decline≥40% | 5 year

SECONDARY OUTCOMES:
Acute coronary syndrome | 5 year
Heart failure | 5 year
Cerebral stroke | 5 year
Peripheral arterial disease | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: xiangmei chen, Principal Investigator — Chinese PLA General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liang S, Wang WL, Zhu FL, Duan SW, Sun XF, Chen XM, Cai GY; Chinese observational prospective study of ageing population with chronic kidney disease (C-OPTION). Chinese observational prospective study of ageing population with chronic kidney disease (C-OPTION): a study protocol. BMJ Open. 2018 Feb 24;8(2):e019457. doi: 10.1136/bmjopen-2017-019457. PMID 29478020